CLINICAL TRIAL: NCT02685878
Title: Physical, Psychological, and Reproductive Outcomes of Women After Obstetric Fistula Repair
Brief Title: Outcomes of Women After Obstetric Fistula Repair
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: UNCPM 21502
Record Dates: First submitted 2016-01-22; First posted 2016-02-19 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Fistula; HIV
Keywords: urinary continence; prevalence of depression; reproductive outcomes; quality of life; HIV status; obstetric fistula
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the long-term surgical success, quality of life, prevalence of depression, fertility rates, and pregnancy outcomes of patients who have undergone obstetric fistula repair.

This will be a study involving up to 300 women 1-3 years after they have undergone obstetric fistula repair at the Fistula Care Center in Lilongwe, Malawi.

Patients who underwent obstetric fistula repair between January 1, 2012 and July 31, 2014 will be identified from an existing database of fistula patients. They will then be contacted and invited to participate in the study. Consented patients will complete a 1-hour pad weight to evaluate urinary continence, a demographic questionnaire, an incontinence-related quality of life metric, and a depression metric. The data will be analyzed and then disseminated to stakeholders.

DETAILED DESCRIPTION:
Eligible participants will be identified from an existing, secure database. Participants will be contacted and traced. They will then be invited to participate in the study. If a participant agrees to participate in the study, they will undergo informed consent by trained study staff, using IRB-approved informed consent forms. They will then undergo a 1-hour pad weight, complete demographic data, complete an incontinence-related quality of life metric, and complete a depression metric.

1-hour pad weight: Use of the 1-hour pad weights have been recommended as an objective measure of treatment outcome for anti-incontinence procedures. After a woman has agreed to enroll in the study and has given written consent, she will be asked to complete a 1-hour pad weight. Pad weights will be measured through having participants sit on a pre-weighed pad for exactly one hour and re-weighing the same pad. The weight of the pad before and after will be recorded and the difference between the two will be used as the pad weight. The pad weight represents the degree of urinary leakage a woman is experiencing. In continent populations, this weight is <1.5 grams. The research assistant will use a calibrated portable scale and stopwatch to ensure accurate recording of these weights. During this time, the remainder of the survey will be conducted.

Demographic Data: Demographic data for each participant will be collected at the time of enrollment and after a written consent has been obtained. This includes information about the patient's age, place of residence, HIV status, education attainment, living arrangement, number of pregnancies and living children, and symptoms of urinary or fecal leakage.

Incontinence-related Quality of Life Metric: To assess OF repair success and continence, participants will be asked about any leakage symptoms with the Kings' Health Questionnaire.

Depression Metric:The 9-question Patient Health Questionnaire (PHQ-9) will be used to assess repaired OF participants for depression.

ELIGIBILITY:
Inclusion Criteria:

1. Study participants who have had an obstetric fistula repair performed at the Fistula Care Center between January 1, 2012 and July 31, 2014
2. Women that currently reside within the districts of Lilongwe, Dedza, Kasungu, Salima, Dowa, Ntcheu, Nkhotakota, Mchinji, Ntchisi, and Mzimba will be traced.
3. Ability to speak Chichewa or English fluently
4. Current age 18 years or above

Exclusion Criteria:

1. Participants who did not have an obstetric fistula repair
2. Participants who have deceased since their obstetric fistula repair
3. Participants who do not currently reside within the districts of Lilongwe, Dedza, Kasungu, Salima, Dowa, Ntcheu, Nkhotakota, Mchinji, Ntchisi, and Mzimba

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 women 1-3 years after they have undergone obstetric fistula repair at the Fistula Care Center in Lilongwe, Malawi.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
The prevalence of participants with a 1-hour pad weight over 1.5 grams (marker of incontinence) will be be calculated. | 1 hour
  To assess OF repair success and continence, patients will complete a 1-hour pad weight, which correlates to urinary incontinence.

SECONDARY OUTCOMES:
Depression after obstetric fistula repair | 1-3 years after obstetric fistula repair
  The PHQ-9 will be administered and women who score a 10 or greater will be considered to have major depression.

OTHER OUTCOMES:
Number of fertile women able to achieve pregnancy after fistula repair | 1-3 years after obstetric fistula repair
  The number of women with any pregnancy since repair divided by the number of married, fecund women.
Quality of life of women after fistula repair | 1-3 years after obstetric fistula repair
  The number of women with a score over 0 in the each of the following domains of the King's Health Questionnaire: general health, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, and sleep/energy.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tang, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Project, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kopp DM, Wilkinson J, Bengtson A, Chipungu E, Pope RJ, Moyo M, Tang JH. Fertility outcomes following obstetric fistula repair: a prospective cohort study. Reprod Health. 2017 Nov 28;14(1):159. doi: 10.1186/s12978-017-0415-1. PMID 29179770